CLINICAL TRIAL: NCT03555292
Title: Safety and Diagnostic Performance of 11C-PIB PET/CT in Patients With Parkinson's Disease and Parkinsonian Dementia Syndromes
Brief Title: 11C-PIB PET/CT in Patients With Parkinson's Disease and Parkinsonian Dementia Syndromes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oriental Neurosurgery Evidence-Based-Study Team (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CPBD2018
Record Dates: First submitted 2018-04-24; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
Keywords: 11C-PIB; Parkinson's disease; dementia; mild cognitive impairment
MeSH Terms: conditions — Parkinson Disease; Dementia; Cognitive Dysfunction | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PD without dementia (Experimental): 11C-PIB injection and PET/CT scan The subjects were intravenously injected with 555MBq 11C-PIB and underwent PET/CT scan immediately after the injection.
  Interventions: Drug: 11C-PiB
- PD with MCI (Experimental): 11C-PIB injection and PET/CT scan The subjects were intravenously injected with 555MBq 11C-PIB and underwent PET/CT scan immediately after the injection.
  Interventions: Drug: 11C-PiB
- PD with dementia (Experimental): 11C-PIB injection and PET/CT scan The subjects were intravenously injected with 555MBq 11C-PIB and underwent PET/CT scan immediately after the injection.
  Interventions: Drug: 11C-PiB
- dementia with Lewy bodies (Experimental): 11C-PIB injection and PET/CT scan The subjects were intravenously injected with 555MBq 11C-PIB and underwent PET/CT scan immediately after the injection.
  Interventions: Drug: 11C-PiB
- healthy control (Experimental): 11C-PIB injection and PET/CT scan The subjects were intravenously injected with 555MBq 11C-PIB and underwent PET/CT scan immediately after the injection.
  Interventions: Drug: 11C-PiB

INTERVENTIONS:
Drug: 11C-PiB — 11C-PIB with 555MBq were intravenously injected into the patients immediately before the PET/CT scans

SUMMARY:
To evaluate the potential contribution of amyloid burden, as indexed by 11C-Pittsburgh compound B (PiB) retention, to the progression of cognitive impairments in patients with Parkinson's disease(PD).

DETAILED DESCRIPTION:
Study design:

Multi-center, Five-arm

Subjects:

Patients with PD without dementia; Patients with PD with mild cognitive impairment (MCI); Patients with PD with dementia; Patients with a dementia with Lewy bodies(DLB); Healthy person

Sample size:

200, including a PD without dementia group of 75 patients, a PD with MCI group of 30 patients, a PD with dementia group of 20 patients, a DLB group of 25 patients and a normal control group of 50 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Parkinson's disease and parkinsonian dementia syndromes
2. Males and females, ≥40 years old
3. The diagnosis of PD is established using the UK Parkinson's Disease Society Brain Bank Research Center Clinical diagnostic criteria. Criteria for PD-MCI and PD-dementia are consistent with those of the Movement Disorder Society. The DLB Consortium consensus criteria are used for DLB.
4. They rely on a combination of neurologic examination and neuropsychological assessment with a battery of tests. Clinical diagnosis was established by sophisticated neurologists.

Exclusion Criteria:

1. Females planning to bear a child recently or with childbearing potential
2. Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
3. Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
4. Known severe allergy or hypersensitivity to IV radiographic contrast.
5. Patients not able to enter the bore of the PET/CT scanner.
6. Inability to lie still for the entire imaging time because of cough, pain, etc.
7. Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
8. Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2021-05-12 (Estimated); Study Completion 2021-10-12 (Estimated)

PRIMARY OUTCOMES:
Amyloid burden range in all subjects | 1 week
  Outcome Measures: All patients underwent a 90-min dynamic 11C-PIB PET scan. 11C-PiB distribution volume ratio (DVR) will be estimated by using the PMOD software.

SECONDARY OUTCOMES:
The cognitive scores in all patients | 0, 6month, 1year
  Functional status is assessed by the Mini-Mental State Examination (MMSE). Parkinson disease with mild cognitive impairment：MMSE score 24-28; Parkinson disease with dementia: MMSE score ≤24; Parkinson disease with normal cognition: MMSE score >28.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Gao, MD, Study Director — Tianjin Medical University General Hospital
Locations (3):
- China (3):
  - Peking Tian Tan Hospital, Capital Medical University, Beijing
  - Tianjin Huanhu Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin